CLINICAL TRIAL: NCT00518752
Title: Comprehensive Oral Care for the Intubated Neuroscience ICU Patient: A Comparison of the Safety and Efficacy Between 2 Protocols
Brief Title: Effects of Oral Care in the Neuroscience ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07NU018-1
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Ventilator Associated Pneumonia; Oral Hygiene
Keywords: Ventilator Acquired Pneumonia; Oral Hygiene; Oral Care; Xerostomia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Xerostomia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Standard Oral Care
  Interventions: Procedure: Standard Oral Care
- B (Experimental): Comprehensive Oral Care
  Interventions: Procedure: Comprehensive Oral Care

INTERVENTIONS:
Procedure: Standard Oral Care — Patients in this arm will receive standard oral care with manual brushes and routine oral hygiene products twice a day
  Arms: A
Procedure: Comprehensive Oral Care — Patients will receive a comprehensive oral care protocol using mechanical brushes and oral care products formulated for patients with a dry mouth twice a day
  Arms: B

SUMMARY:
The purpose of this study is to compare how effective different ways of mouth cleaning are for patients in a neuroscience intensive care unit with a breathing tube in their mouth.

DETAILED DESCRIPTION:
Patients with neurological dysfunction requiring intubation and ventilation are at risk for developing ventilator acquired pneumonia. Several studies have suggested that oral hygiene plays a role in the subsequent development of pneumonia for patients in the intensive care unit requiring intubation and mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* > or equal 18 years old
* Intubated within 24hours of admission to the Neuroscience ICU
* Intubation anticipated to continue for approximately 72 hours

Exclusion Criteria:

* Minors
* Pregnancy
* Acute cervical spinal cord injury
* Severe facial trauma
* Family not present for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2007-05; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Development of Ventilator Acquired Pneumonia | During the period of intubation

SECONDARY OUTCOMES:
Improved Oral Health | During the period of intubation and 48 hours following extubation

CONTACTS AND LOCATIONS:
Overall Officials: Virginia C Prendergast, MSN, NP-C, Principal Investigator — St Joseph's Hospital and Medical Center, Phoenix, Arizona, USA; Ingalill R Hallberg, PhD, Study Chair — Vardalinstitutet, University of Lund, Sweden
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Background] Munro CL, Grap MJ. Oral health and care in the intensive care unit: state of the science. Am J Crit Care. 2004 Jan;13(1):25-33; discussion 34. PMID 14735645
- [Background] Dennesen P, van der Ven A, Vlasveld M, Lokker L, Ramsay G, Kessels A, van den Keijbus P, van Nieuw Amerongen A, Veerman E. Inadequate salivary flow and poor oral mucosal status in intubated intensive care unit patients. Crit Care Med. 2003 Mar;31(3):781-6. doi: 10.1097/01.CCM.0000053646.04085.29. PMID 12626984
- [Derived] Prendergast V, Hagell P, Hallberg IR. Electric versus manual tooth brushing among neuroscience ICU patients: is it safe? Neurocrit Care. 2011 Apr;14(2):281-6. doi: 10.1007/s12028-011-9502-2. PMID 21249529